CLINICAL TRIAL: NCT06719024
Title: A Randomized Controlled Trial to Assess the Efficacy and Safety of Topical Ruxolitinib for Face and Neck Vitiligo of Adult Chinese Patients Refractory to Topical Tacrolimus
Brief Title: Topical Ruxolitinib for Face and Neck Vitiligo of Adult Chinese Patients Refractory to Topical Tacrolimus
Acronym: RCT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Yuk Ming Lau, Principal Investigator, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-613
Record Dates: First submitted 2024-11-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Vitiligo
Keywords: non-segmental vitiligo; randomized controlled trial; Chinese
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ruxolitinib cream (Active Comparator): a thin layer of the assigned topical to the selected lesions twice daily
  Interventions: Drug: Ruxolitinib Cream 1.5%
- Aqueous cream (Placebo Comparator): a thin layer of the assigned topical to the selected lesions twice daily
  Interventions: Drug: Aqueous cream

INTERVENTIONS:
Drug: Ruxolitinib Cream 1.5% — a thin layer of the assigned topical to the selected lesions twice daily, maintaining at least an 8-hour interval between applications
  Arms: Ruxolitinib cream
Drug: Aqueous cream — a thin layer of the assigned topical to the selected lesions twice daily, maintaining at least an 8-hour interval between applications
  Arms: Aqueous cream

SUMMARY:
This trial is a prospective, open-label, single-center, split face randomized controlled study comparing 1.5% topical Ruxolitinib cream twice daily (BD) to aqueous cream in treating non-segmental vitiligo (NSV) of the face and neck in patient previous failed to respond to topical tacrolimus 0.1%. Aqueous cream twice daily application will be used as control group treatment. Patients with stable NSV at least 0.5% of their total body surface area (BSA) on the face and neck, as determined by the fingertip method, are screened. Recruited subjects will be asked to review their impression of change of their lesion by the end of the study using a 7-point scale.

DETAILED DESCRIPTION:
Vitiligo is a chronic autoimmune skin disorder marked by the loss of melanocytes, leading to the development of depigmented patches on the skin. In this study, the investigators hypothesis that there is a noticeable difference in responses between using 1.5% ruxolitinib cream applied twice daily (BD) and aqueous cream BD at the end of the trial period. The investigators aim to investigate the efficacy and safety of topical 1.5% topical ruxolitinib cream on non-segmental vitiligo of the face and neck in Chinese patients who previously failed to improve with topical tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 year old
* Have a clinical diagnosis of stable non-segmental vitiligo
* Depigmentation including at least 0.5% of the BSA on the face and neck
* Previously treated with topical tacrolimus 0.1% BD for at least 3 months without significant response
* Agree to stop using any topical treatments on face and neck and systemic treatment for vitiligo during the washout period until the trial concludes. Use of over-the-counter products approved by the investigator and camouflage makeup is allowed
* Both male and female patients must commit to using effective birth control to prevent pregnancy or fathering a child throughout the study
* Subjects or their legally authorized representative, if applicable, must be able to understand and willing to provide informed consent at Screening visit

Exclusion Criteria:

* Patients who refuse to give consent
* Presence of different vitiligo types or other skin depigmentation conditions like piebaldism or leprosy, etc.
* History of using depigmentation treatments other than hydroquinone for vitiligo or pigmentation issues
* Any skin condition affecting study participation, active skin infections one week before the study starts, issues impacting vitiligo evaluation, or serious health problems limiting involvement or increasing risk
* Significant medical disease that may hinder use of topical JAK inhibitor, e.g. serious infection, untreated chronic hepatitis, malignancy within 5 years except adequately treated non metastatic cancer, evidence of clinically significant or uncontrolled cardiovascular disease, thrombosis including DVT and PE, blood abnormality including significant thrombocytopenia, anaemia (Hb <10g/dL) and significant neutropenia, substance misuse
* Specific treatment use within certain periods before starting (Baseline visit):

  1 week for topical vitiligo treatments 4 weeks for immunomodulators, photosensitizers, oral retinoids, methoxsalen, or live vaccines 8 weeks for laser or phototherapy on face and neck 12 weeks for biologics
* Any prior application of topical or oral JAK inhibitors
* Hemoglobin under 10 g/dL, significant liver dysfunction, and/or evidence of HIV infection or positive for HIV antibodies at initial screening or current acquired, common variable or inherited, primary or secondary immunodeficiency
* Females of childbearing potential who are pregnant, during breastfeeding period, or those planning pregnancy during the study
* Those unlikely or unable to comply with the requirements of this study protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Degree of repigmentation at week 24 comparing to baseline | week 24
  Comparing the degree of repigmentation of lesion site between baseline and week 24 with Physician global assessment of the degrees of repigmentation of the vitiligo lesions

CONTACTS AND LOCATIONS:
Overall Officials: YM Lau, Principal Investigator — Queen Mary Hospital, Hospital Authority
Locations (1):
- Queen Mary Hospital, Hospital Authority, Hong Kong, Hong Kong